CLINICAL TRIAL: NCT00766818
Title: The Effect of Pregnancy on the Pharmacokinetics of the Kaletra Tablet: A Longitudinal Investigation in the Second and Third Trimesters Including Empiric Dosage Adjustment
Brief Title: The Effect of Pregnancy on the Pharmacokinetics of the Kaletra Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Angela Kashuba, PharmD, University of North Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #06-0653
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy; HIV
MeSH Terms: interventions — lopinavir-ritonavir drug combination; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Kaletra
  Interventions: Drug: Kaletra

INTERVENTIONS:
Drug: Kaletra — Kaletra 400/100mg BID, then increase at 30weeks to 500/125mg BID
  Other Names: lopinavir; ritonovir

SUMMARY:
In this study, we are looking at blood concentrations of Kaletra in HIV positive patients during pregnancy. The patients will come in for 4 visits lasting ~24hrs. These visits take place at 20-24 weeks, 30 weeks, 32 weeks and 8 weeks post-partum. At the end of vist 2 (week 30), we will increase your dose to 2 adult Kaletra tablets, and one pediatric Kaletra tablet (total dose 500/125mg). The dose will remain increased until you are 2 weeks post partum, then it will return to the standard 2 adult tablets (400/100mg).

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Pregnant (<22 weeks)
* Currently taking or planning to start Kaletra
* ≥18 years of age

Exclusion Criteria:

* Active opportunistic or serious bacterial infection at the time of entry
* Past or present obstetrical complications (including, but not limited to: placentia previa, eclampsia, confirmed birth defects, multiple gestation pregnancies)
* Unable to maintain medication adherence, defined as ≥ 80% of doses taken between visits
* Currently receiving or expected to receive other protease inhibitors in conjunction with Kaletra®
* HIV genotype showing accumulation of protease inhibitor mutations expected to result in virologic failure on Kaletra® OR documented virologic failure on Kaletra®-containing regimen attributable to the Kaletra® component
* Chronic hepatitis B and/or C virus infection
* Cushing's Syndrome
* Untreated hypothyroidism or hyperthyroidism
* Serum Creatinine > 1.5 mg/dL
* Amylase 1.5 times ULN and/or abnormal lipase
* Direct or total bilirubin levels > Grade 1
* ALT/AST > Grade 2 (based on the NIH Division of AIDS (DAIDS) Table for Grading the Severity of Adverse Events
* Bicarbonate > Grade 2 (DAIDS)
* Hematology > Grade 2 (DAIDS), except for anemia: exclude only women with Hb< 9 g/dL and/or HCT , 27.3% (< 8.5 mg/dL and/or HCT , 25.6% if currently on ZDV) at screening; all subjects with anemia who enroll in the study must be receiving or start hematinics, including iron and folate supplements, immediately upon enrollment and continue until anemia resolves or end of pregnancy. The hematinic supplements may be discontinued at the discretion of the investigator if they consider continuation would not be in the best interest of the subject.
* Receiving the following drugs: astemizole, terfenadine, rifampin, cisapride, ergot derivatives, simvastatin, lovastatin, St. John's wort, pimozide, midazolam, triazolam, carbamezapine, phenobarbital, phenytoin, or dexamethasone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To compare the C12h and AUC0-12h of protein bound and unbound blood plasma lopinavir (LPV) using standard doses during the second and third trimesters of pregnancy. | 20-24 weeks, 30weeks, 32 weeks gestation and 8 weeks postpartum
To compare the C12h and AUC0-12h of protein bound and unbound blood plasma LPV between standard doses (400mg/100mg BID) and increased doses (500/125mg BID) of Kaletra® during the third trimester of pregnancy. | 20-24weeks, 30 weeks, 32 weeks gestation, 8weeks postpartum

SECONDARY OUTCOMES:
To compare the C12h and AUC0-12h of protein bound and unbound blood plasma ritonavir (RTV) using standard doses during the second and third trimesters of pregnancy. | 20-24weeks, 30weeks, 32weeks gestation, 8 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina; Kristine B Patterson, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States